CLINICAL TRIAL: NCT06031376
Title: Fruquintinib With PD-1 Inhibitors Versus TAS-102 With Bevacizumab in Late-Line mCRC: A Retrospective Cohort Study Based on Propensity Score Matching
Brief Title: Fruquintinib With PD-1 Inhibitors Versus TAS-102 With Bevacizumab in Late-Line mCRC
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FPTB-01
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: Colorectal cancer; Fruquintinib;PD-1;TAS-102; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013; Immune Checkpoint Inhibitors; trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fruquintinib plus PD-1 inhibitors: In fruquintinib plus PD-1 inhibitors group,The patients were treated orally with Fruquintinib (5mg once daily for 14 days on/7 days off, over a 21-day cycle), combined with 1 of the 5 anti-PD-1 antibodies (i.e., nivolumab, pembrolizumab, camrelizumab, sintilimab, or toripalimab). The anti-PD-1 antibody was administered intravenously on day 1, and its recommended dosage was as follows: nivolumab: 240 mg, every 2 weeks; pembrolizumab, camrelizumab, and sintilimab: 200 mg every 3 weeks; and toripalimab: 240 mg every 3 weeks.
  Interventions: Drug: Fruquintinib; Drug: PD-1 inhibitors
- TAS-102 plus bevacizumab: In TAS-102 plus BEV group, Patients received TAS-102 (35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days) and bevacizumab (5 mg /kg, intravenously, on days 1 and 15, every 28 days). Bevacizumab was approved to be a 30-minute intravenous infusion before TAS-102.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Fruquintinib — 5mg once daily for 14 days on/7 days off, over a 21-day cycle
  Groups: Fruquintinib plus PD-1 inhibitors
Drug: PD-1 inhibitors — The anti-PD-1 antibody was administered intravenously on day 1, and its recommended dosage was as follows: nivolumab: 240 mg, every 2 weeks; pembrolizumab, camrelizumab, and sintilimab: 200 mg every 3 weeks; and toripalimab: 240 mg every 3 weeks.
  Other Names: anti-PD-1 antibodies
  Groups: Fruquintinib plus PD-1 inhibitors
Drug: Trifluridine/Tipiracil — TAS-102 35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days
  Other Names: TAS-102; Lonsurf; S 95005
  Groups: TAS-102 plus bevacizumab
Drug: Bevacizumab — Bevacizumab 5 mg /kg, intravenously on days 1,15,every 28 days
  Other Names: Avastin
  Groups: TAS-102 plus bevacizumab

SUMMARY:
Fruquintinib with PD-1 inhibitors (FP) and TAS-102 with bevacizumab (TB) are two common therapies for patients with previous-treated metastatic colorectal cancer (mCRC). However, it's still not clear that which therapy can bring better prognosis. Our study sought to investigate the efficacy and safety of fruquintinib with PD-1 Inhibitors versus TAS-102 with bevacizumab in Late-Line mCRC between July 2019 to October 2022July 2019 and June 2021 at the Hunan Cancer Hospital.

DETAILED DESCRIPTION:
This is a retrospective cohort study conducted in Hunan Cancer Hospital. Patients (pts) with mCRC who had received at least the 2nd line treatment were eligible. Propensity score (PS) would be calculated to balance the baseline characteristics of two arms. Overall survival (OS) was set as the primary endpoint. From July 2019 to October 2022, 106 eligible pts in total were enrolled. According to the treatment received, 72 and 34 pts were respectively allocated into FP cohort and TB cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded).
2. Have progressed from at least 2 lines of standard treatment,including fluoropyrimidines, irinotecan, oxaliplatin, with or without targeted drugs, like bevacizumab and cetuximab (only for RAS wild-type). Regorafenib was permitted but not required for inclusion.
3. Has measurable or non-measurable disease as defined by RECIST version 1.1
4. Is able to swallow oral tablets.
5. Estimated life expectancy ≥12 weeks.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) less than 2
7. Has adequate organ function.

Exclusion Criteria:

1. Pregnancy, lactating female or possibility of becoming pregnant during the study.
2. Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy (excluding alopecia, and skin pigmentation).
3. Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.
4. Has severe or uncontrolled active acute or chronic infection.
5. Known carriers of HIV antibodies.
6. Confirmed uncontrolled arterial hypertension or uncontrolled or symptomatic arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population were the patients treated with at least 2 cycle of fruquintinib plus PD-1 Inhibitors or TAS-102 plus BEV in patients suffering refractory mCRC from July 2019 to October 2022 at the Hunan Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of commencement of treatment and the date of death due to any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the date of commencement of treatment and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.
Overall response rate (ORR) | Approximately 12 months
  Overall response rate (ORR) was regarded as the proportion of complete responses (CRs) and partial responses (PRs) according to RECIST version 1.1 criteria and using investigator's tumor assessment
Disease control rate (DCR) | Approximately 12 months
  Disease control rate has been defined as the addition of (CR + PR) rate and also stable disease (SD) rate
Treatment-Related Adverse Events (TRAE) | Approximately 12 months
  Treatment-Related Adverse Events (TRAE) as assessed by CTCAE v5.0, including serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Rongrong li, professor, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for principal investigator or correspondence author]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author.